CLINICAL TRIAL: NCT06682442
Title: Induction Chemotherapy Response-Guided Radiation for EBV-Associated Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24726; NCI-2024-08983 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Nasopharyngeal Carcinoma; Stage III Nasopharyngeal Carcinoma AJCC v8; Stage IVA Nasopharyngeal Carcinoma AJCC v8; Nasopharyngeal Cancer; Nasopharyngeal Cancer Stage
Keywords: HHV-4 Positive; EBV Positive; human herpesvirus 4 (HHV-4) positive
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections | interventions — Radiotherapy, Intensity-Modulated; Phantoms, Imaging; Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (de-escalated Intensity Modulated Radiation Therapy (IMRT) (Experimental): Participants undergo de-escalated IMRT every day (QD) 5 days a week for up to 7 weeks in the absence of disease progression or unacceptable toxicity. Participants also undergo CT, MRI, PET, PET/CT, CT, and/or bone scans as well as providing blood samples throughout the trial.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy (IMRT); Procedure: Radiographic Imaging; Procedure: Biospecimen Collection
- Arm II (standard IMRT) (Experimental): Patients undergo standard IMRT QD 5 days a week for up to 7 weeks in the absence of disease progression or unacceptable toxicity. Participants also undergo CT, MRI, PET, PET/CT, CT, and/or bone scans as well as providing blood samples throughout the trial.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy (IMRT); Procedure: Radiographic Imaging; Procedure: Biospecimen Collection

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT
Procedure: Radiographic Imaging — Undergo imaging procedure
  Other Names: PET Scan; Positron Emission Tomography (PET); Computed Tomography (CT); CT; Magnetic Resonance Imaging (MRI); MRI; PET MRI; PET CT
Procedure: Biospecimen Collection — Blood samples will be collected
  Other Names: Blood Specimen; Blood Sample

SUMMARY:
This clinical trial tests the effect of induction chemotherapy response-guided radiation (de-escalated intensity-modulated radiation therapy [IMRT]) compared to standard IMRT in patients with Epstein-Barr virus (EBV)-associated nasopharyngeal cancer. Intensity-modulated radiation therapy (IMRT) is an advanced form of 3-dimensional radiation therapy that uses computer-generated images to show the size and shape of the tumor. Thin beams of radiation of different intensities are aimed at the tumor from many angles. This type of radiation therapy reduces the damage to healthy tissue near the tumor. Radiation therapy sometimes causes unwanted symptoms or side effects, including late effects such as hearing loss and dental problems. The severity of the side effects is related to the radiation dose received and the amount of tissue that received radiation. De-escalation IMRT uses lower doses of radiation based on a good response to induction chemotherapy. Giving de-escalated IMRT may be as effective as standard doses of IMRT in treating patients with EBV-associated nasopharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To measure the proportion of participants alive without progression of disease two years following induction therapy (IT) response-guided IMRT.

SECONDARY OBJECTIVES:

I. To assess the 1-year rate of progression-free survival (PFS) after IT response-guided IMRT.

II. To assess the 1- and 2-year cumulative incidence of locoregional recurrence (LRR) after IT response-guided IMRT.

III. To assess the 1- and 2-year cumulative incidence of distant metastasis (DM) after IT response-guided IMRT.

IV. To assess the 1- and 2-year rates of overall survival (OS) after IT response-guided IMRT.

V. To compare the rates of severe acute toxicities between standard and de-escalated IMRT.

VI. To compare the rates of severe late toxicities between standard and response-guided IMRT over a period of 2 years.

EXPLORATORY OBJECTIVES:

I. To compare the frequency of radiation treatment breaks between standard and de-escalated IMRT.

II. To compare the frequency of hospitalizations between standard and de-escalated IMRT.

III. To compare pre-treatment and short- and long-term post-treatment quality of life (QoL) after standard versus de-escalated IMRT.

IV. To compare pre-treatment and short- and long-term post-treatment levels of fatigue after standard versus de-escalated IMRT.

V. To compare radiation dosimetric parameters between standard and de-escalated IMRT.

VI. To explore differences in efficacy endpoints by sex, age, English language status, and race/ethnicity.

VII. To explore heterogeneity of treatment effects (HTEs) of efficacy endpoints by variables, such as sex, age, English language status, and race/ethnicity.

VIII. To explore the association between EBV deoxyribonucleic acid (DNA) levels and disease response on imaging upon completion of IT.

IX. To explore longitudinal EBV DNA levels after completion of IT response-guided IMRT.

X. To compare the rates of severe very late toxicities (from years 2 to 10 after completion of IMRT) between standard and response-guided IMRT.

XI. To explore the association between adjuvant (post-chemoradiation) systemic therapy use and oncologic outcomes (PFS, locoregional recurrence, distant metastasis, and overall survival), quality of life, and fatigue.

XII. To assess frequency of intra-treatment tumor hypoxia in participants undergoing standard and de-escalated radiotherapy.

XII. To explore the association between the presence of intra-treatment tumor hypoxia and baseline demographic and clinical characteristics.

XIV. To explore the association between the presence of intra-treatment tumor hypoxia and oncologic outcomes, toxicity, quality of life, and fatigue.

XV. To evaluate the relationship between intra-treatment tumor hypoxia and pre-treatment EBV DNA levels.

XVI. To evaluate the relationship between intra-treatment tumor hypoxia and end-of-treatment EBV DNA levels.

OUTLINE: Patients with partial radiographic response to IT in the primary tumor and lymph nodes are assigned to Arm I. Patients with stable or progressive disease are assigned to Arm II.

ARM I (DE-ESCALATED INTENSITY): Patients undergo de-escalated IMRT once daily (QD) 5 days a week for up to 7 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT)/magnetic resonance imaging (MRI), positron emission tomography (PET), PET/CT, CT, and/or bone scans throughout the trial

ARM II (STANDARD): Patients undergo standard IMRT QD on 5 days a week for up to 7 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT/MRI, PET, PET/CT, CT, and/or bone scans throughout the trial.

After completion of study treatment, patients are followed up at 3 months then every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed (from primary lesion and/or lymph nodes) nasopharyngeal carcinoma.
* Participants must have Epstein Barr virus (EBV)-associated nasopharyngeal carcinoma, defined as detectable (> 0 copies/mL) circulating plasma EBV DNA on a qualitative or quantitative polymerase chain reaction (PCR)-based test.
* Stage III-IVA disease (American Joint Committee on Cancer [AJCC], 8th edition [ed.]) with no evidence of distant metastasis at the time of diagnosis based upon all 3 of the following minimum diagnostic workup criteria:

  * History/physical examination by a medical oncologist or clinical oncologist or radiation oncologist or otolaryngology (ENT);
  * Evaluation of tumor extent with either one of the following:

    * MRI with contrast of the face, nasopharynx, and neck or CT with contrast of the face, nasopharynx and neck with ≤ 3 mm contiguous slices and bone windows to evaluate base of skull involvement; or
    * MRI of the nasopharynx and PET/CT (with contrast) of the neck
  * Imaging to rule out distant metastasis:

    * CT scan with contrast of the chest and abdomen (required) and the pelvis (optional) or a total body PET/CT scan (non-contrast PET/CT is acceptable); and
    * Only if clinically indicated: Bone scan only when there is suspicion of bone metastases (a PET/CT scan can substitute for the bone scan)
* Started or planning to start platinum-based induction systemic therapy.
* Planning to receive intensity modulated radiation therapy (IMRT) with concurrent, platinum-based systemic therapy during radiation.
* Use of adjuvant (post-chemoradiation) immunotherapy is permitted.
* Age >=18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 50%).
* Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy are eligible for this trial.
* For individuals with evidence of chronic hepatitis B virus (HBV) infection: must be on suppressive therapy, if indicated.
* For individuals with a history of hepatitis C virus (HCV) infection: must be currently on treatment, or must have been treated and cured.
* Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Because the radiation therapy used in this trial is known to be teratogenic, individuals of reproductive potential must agree to use adequate contraception (e.g., hormonal or barrier methods, abstinence) for the duration of study participation and for at least 60 days after the last administration of radiation therapy. Should a study participant or their partner become pregnant or suspect pregnancy while participating in this study, they should inform their treating physician immediately.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior systemic chemotherapy for nasopharyngeal carcinoma, other than induction chemotherapy (IT); note that prior chemotherapy for a different cancer is permitted
* Prior radiotherapy to the nasopharynx or surrounding involved areas that would result in overlap of radiation therapy fields
* Has participated in a study of an investigational product and received treatment with an investigational drug or used an investigational device within 4 weeks prior to the first dose of treatment
* Severe, active comorbidity, defined as any of the following:

  * Major medical or psychiatric illness that, in the treating investigator's opinion, would interfere with the completion of therapy and follow-up or interfere with a full understanding of the risks and potential complications of the therapy
  * Unstable angina, congestive heart failure, or peripheral vascular disease requiring hospitalization within the last 12 months; or other cardiac compromise that in the judgment of the treating investigator will preclude safe administration of study treatment
  * Chronic obstructive pulmonary disease (COPD) exacerbation or other respiratory illness requiring hospitalization within 30 days prior to registration, or which would preclude safe administration study therapy in the opinion of the treating investigator
  * Active, untreated infection and/or acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Because the radiation therapy used in this trial is known to be teratogenic, individuals of child-bearing potential must have documentation in their medical record of a negative pregnancy test

  * A female participant is considered to NOT be of child-bearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), if the participant meets either of the following two criteria:
  * Has reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause)
  * Has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries)
* Individuals with any condition or social circumstance that, in the opinion of the investigator, would impair the participant's ability to comply with study activities or interfere with participant safety or study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival Rate (PFS) at 2 years post radiation | Up to 26 months
  PFS is defined as the proportion of participants alive without progression of disease from the first day of radiotherapy to progression or death by any cause, whichever occurs first, assessed up to 2 years after the last day of radiation therapy. The Kaplan-Meier method will be used to estimate the PFS rate along with a 90% confidence interval.

SECONDARY OUTCOMES:
Progression-Free Survival Rate (PFS) at 1 year post radiation | Up to 14 months
  PFS is defined as the proportion of participants alive without progression of disease from the first day of radiotherapy to progression or death by any cause, whichever occurs first, assessed up to 1 year after the last day of radiation therapy. The Kaplan-Meier method will be used to estimate the PFS rate along with a 90% confidence interval.
Locoregional recurrence rate (LRR) at 1 year post radiation | Up to 14 months
  LRR will be estimated using cumulative incidence from the first day of radiation to 1 year after the last day of radiation.
Locoregional recurrence rate (LRR) at 2 years post radiation | Up to 26 months
  LRR will be estimated using cumulative incidence from the first day of radiation to 2 years after the last day of radiation.
Incidence of Distant metastasis (DM) at 1 year post radiation | Up to 14 months
  DM will be estimated using cumulative incidence from the first day of radiation to 1 year after the last day of radiation.
Incidence of Distant metastasis (DM) at 2 years post radiation | Up to 26 months
  DM will be estimated using cumulative incidence from the first day of radiation to 2 years after the last day of radiation.
Median Overall Survival (OS) at 1 year post radiation | Up to 14 months
  Kaplan-Meier will be used to estimate OS
Median Overall Survival (OS) at 2 years post radiation | Up to 26 months
  Kaplan-Meier will be used to estimate OS
Overall Proportion of patients with grade ≥ 3 adverse events (AEs) | Up to 5 months
  Adverse Events will be reported from the start of radiation until 3 months after completion of radiation and will be graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The percent of participants will be reported overall.
Proportion of patients with acute grade ≥ 3 adverse events (AEs) by group | Up to 5 months
  Any adverse events from the start of radiation until 3 months after completion of radiation with a grade 3 or higher as determined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 will be reported as a percentage of the total participants for each treatment group.
Proportion of patients with late onset grade ≥ 3 AEs by group post radiation | Up to 21 months
  Any adverse events from 3 months after completion radiation until 2 years after completion of radiation, with a grade 3 or higher as determined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 will be reported as a percentage of the total participants for each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Yom, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No